CLINICAL TRIAL: NCT01721161
Title: A Randomized, Double-Blind, Parallel-Group, Placebo Controlled Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of BIIB033 in Subjects With First Episode of Acute Optic Neuritis
Brief Title: BIIB033 In Acute Optic Neuritis (AON)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215ON201
Record Dates: First submitted 2012-10-25; First posted 2012-11-05 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Acute Optic Neuritis
Keywords: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — opicinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIIB033 (Experimental): Participants will receive BIIB033 once every 4 weeks for 20 weeks (a total of 6 doses).
  Interventions: Biological: BIIB033 (anti-LINGO-1 mAb)
- Placebo (Placebo Comparator): Participants will receive Placebo via IV infusion once every 4 weeks for 20 weeks (a total of 6 doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: BIIB033 (anti-LINGO-1 mAb) — 100 mg/kg via IV infusion once every 4 weeks for 20 weeks (a total of 6 doses).
  Other Names: anti-LINGO-1 monoclonal antibody (mAb); Opicinumab
  Arms: BIIB033
Drug: Placebo — via IV infusion once every 4 weeks for 20 weeks (a total of 6 doses)
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of BIIB033 in subjects with their first episode of unilateral acute optic neuritis (AON). The secondary objective of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of BIIB033 in this study population.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to provide written consent and any authorization required by law.
* Confirmed diagnosis of AON
* All male or female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for at least 6 months after their last dose of study treatment.

Key Exclusion Criteria:

* Prior episode(s) of optic neuritis or loss of vision not due to AON.
* Subjects with an established diagnosis of multiple sclerosis are excluded except if newly diagnosed based on the current episode of AON and positive brain magnetic resonance imaging results consistent with the 2010 revisions to the McDonald's criteria.
* Previous history of a clinically significant disease.
* Females who have a positive pregnancy test result, or who are pregnant, breastfeeding, or planning to conceive during the study.
* History of human immunodeficiency virus (HIV), hepatitis C virus antibody, or hepatitis B virus.
* History or evidence of drug or alcohol abuse within 2 years prior to Screening.
* Current enrollment in any other study treatment or disease study within 3 months prior to Day 1/Baseline.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (32):
- Australia (2):
  - Research Site, Parkville
  - Research Site, Sydney
- Belgium (4):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Limbourg
- Canada (2):
  - Research Site, Halifax
  - Research Site, Ottawa
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Glostrup Municipality, Denmark
- Germany (5):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Tübingen
- Research Site, Budapest, Hungary
- Italy (4):
  - Research Site, Fidenza
  - Research Site, Florence
  - Research Site, Milan
  - Research site, Roma
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Palmar
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Lund
  - Research Site, Stockholm
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London

REFERENCES:
- [Derived] Klistorner A, Chai Y, Leocani L, Albrecht P, Aktas O, Butzkueven H, Ziemssen T, Ziemssen F, Frederiksen J, Xu L, Cadavid D; RENEW MF-VEP Investigators. Assessment of Opicinumab in Acute Optic Neuritis Using Multifocal Visual Evoked Potential. CNS Drugs. 2018 Dec;32(12):1159-1171. doi: 10.1007/s40263-018-0575-8. PMID 30267385
- [Derived] Petrillo J, Balcer L, Galetta S, Chai Y, Xu L, Cadavid D. Initial Impairment and Recovery of Vision-Related Functioning in Participants With Acute Optic Neuritis From the RENEW Trial of Opicinumab. J Neuroophthalmol. 2019 Jun;39(2):153-160. doi: 10.1097/WNO.0000000000000697. PMID 30095536
- [Derived] Cadavid D, Balcer L, Galetta S, Aktas O, Ziemssen T, Vanopdenbosch L, Frederiksen J, Skeen M, Jaffe GJ, Butzkueven H, Ziemssen F, Massacesi L, Chai Y, Xu L, Freeman S; RENEW Study Investigators. Safety and efficacy of opicinumab in acute optic neuritis (RENEW): a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2017 Mar;16(3):189-199. doi: 10.1016/S1474-4422(16)30377-5. Epub 2017 Feb 15. PMID 28229892

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo via IV infusion once every 4 weeks for 20 weeks (a total of 6 doses)
- BIIB033: BIIB033 100 mg/kg via IV infusion once every 4 weeks for 20 weeks (a total of 6 doses)
Period: Overall Study
Arm/Group | Placebo | BIIB033
Started | 41 | 41
Completed | 37 | 34
Not Completed | 4 | 7
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIIB033 | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (8.85) | 31.8 (7.17) | 32.1 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 10 | 14 | 24
Days from first AON symptom to first dose [Mean (Standard Deviation); unit: days] — First dose given, on average, 2 weeks after completion of high-dose (1 g daily for 3 to 5 days) IV methylprednisolone treatment.
  days | 24.6 (3.4) | 23.6 (4.0) | 24.1 (3.7)
Days from confirmed AON diagnosis to first dose [Mean (Standard Deviation); unit: days] | 19.2 (4.9) | 18.7 (4.7) | 19.0 (4.8)
Affected eye [Number; unit: participants]
  Right eye | 19 | 25 | 44
  Left eye | 22 | 16 | 38
Criteria for AON diagnosis [Number; unit: participants]
  Decreased visual acuity | 36 | 41 | 77
  Decreased color vision | 30 | 33 | 63
  Relative afferent pupillary defect | 34 | 31 | 65
  Visual field defect | 32 | 37 | 69
  Ocular pain | 31 | 36 | 67
  Not specified | 5 | 4 | 9
AON signs and symptoms at screening or baseline [Number; unit: participants] — Symptoms were not uniformly tested in accordance with a predefined protocol.
  participants
    Visual field defect | 29 | 34 | 63
    Color desaturation | 33 | 32 | 65
    Uhthoff's symptom | 8 | 18 | 26
    Swollen optic disc | 8 | 12 | 20
    Relative afferent pupillary defect | 33 | 30 | 63
FF-VEP conduction block in the affected eye at baseline [Number; unit: participants] — FF-VEP=full-field visual evoked potentials
  participants
    FF-VEP conduction block | 5 | 10 | 15
    No FF-VEP conduction block | 36 | 31 | 67
FF-VEP latency in the fellow eye at baseline [Mean (Standard Deviation); unit: ms] | 101.7 (5.25) | 102.7 (6.4) | 102.2 (5.8)
RGCL/IPL thickness in the affected eye at baseline [Mean (Standard Deviation); unit: microns] — RGCL/IPL=retinal ganglion cell layer/inner plexiform retinal layer. n=38 in the placebo group and n=40 in the anti-LINGO-1 group, total n=78.
  microns | 66.0 (6.9) | 63.8 (7.4) | 64.8 (7.2)
Brain Gd+ lesions before first dose [Mean (Standard Deviation); unit: lesions] — Gd+=gadolinium-enhancing. n=38 in each group, total n=76.
  lesions | 0.5 (1.6) | 0.2 (1.0) | 0.4 (1.4)
Volume of brain T2 lesions before first dose [Mean (Standard Deviation); unit: mL] — n=38 in each group, total n=76.
  mL | 1.09 (1.32) | 1.09 (1.90) | 1.09 (1.63)

OUTCOME MEASURES:

1. Primary Outcome: Change in Full-field Visual Evoked Potential (FF-VEP) Latency at Week 24: Intent-to-treat (ITT) Population
Description: Adjusted mean change in optic nerve conduction velocity (NCV) at Week 24 for the affected eye from the baseline of unaffected fellow eye as determined by FF-VEP. Adjusted for the baseline latency of fellow eye.
Time Frame: Baseline, Week 24
Population: ITT population: all randomized subjects who received at least 1 dose of study treatment (BIIB033 or placebo). Last observation carried forward (LOCF) imputation was used if Week 24 data were missing.
Measure: Mean (Standard Error); unit: msec
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 41 | 41
msec | 20.83 (2.53) | 17.34 (2.53)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; Test type: Superiority or Other; p = 0.3337, ANCOVA; Difference = -3.48, 95% CI 2-sided [-10.61 to 3.65] — Difference is calculated as BIIB033 100 mg/kg - placebo

2. Secondary Outcome: Percentage Change in Spectral-domain Optical Coherence Tomography (SD-OCT) Average Retinal Nerve Fiber Layer (RNFL) Thickness at Week 24: ITT Population
Description: Adjusted mean percentage change in thickness of the RNFL at Week 24 for the affected eye from the baseline of unaffected fellow eye as determined by SD-OCT. Percentage change is calculated as (affected eye - baseline of fellow eye)/baseline of fellow eye*100. Adjusted for the baseline RNFL thickness.
Time Frame: Baseline, Week 24
Population: ITT population: all randomized subjects who received at least 1 dose of study treatment (BIIB033 or placebo) and a valid RNFL assessment at Baseline. LOCF imputation was used if Week 24 data were missing.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 39 | 41
percentage change | -11.77 (2.08) | -15.66 (2.03)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; Test type: Superiority or Other; p = 0.1868, ANCOVA; Difference = -3.89, 95% CI 2-sided [-9.70 to 1.92] — Difference is calculated as BIIB033 100 mg/kg - placebo

3. Secondary Outcome: Percentage Change in SD-OCT Average RNFL Thickness at Week 24: Per-protocol Population
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Per-protocol Population: participants from the ITT population who completed the study, did not miss more than 1 dose of BIIB033 or placebo, and did not receive MS-modifying therapies during the study period, which were prohibited per protocol. LOCF imputation was used if Week 24 data were missing.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 35 | 33
percentage change | -12.22 (2.26) | -16.98 (2.33)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; Test type: Superiority or Other; p = 0.1488, ANCOVA; Difference = -4.76, 95% CI 2-sided [-11.26 to 1.74]

4. Secondary Outcome: Change in SD-OCT Average Retinal Ganglion Cell Layer/Inner Plexiform Retinal Layer (RGCL/IPL) at Week 24: ITT Population
Description: Adjusted mean change in thicknesses of the RGCL/IPL at Week 24 for the affected eye from the baseline of unaffected fellow eye as determined by segmentation of SD-OCT. Adjusted for the baseline RGCL/IPL thickness.
Time Frame: Baseline, Week 24
Population: ITT population: all randomized subjects who received at least 1 dose of study treatment (BIIB033 or placebo) with a valid RGCL/IPL assessment at Baseline. LOCF imputation was used if Week 24 data were missing.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 40 | 41
µm | -9.90 (1.20) | -11.05 (1.18)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; Test type: Superiority or Other; p = 0.4975, ANCOVA; Difference = -1.15, 95% CI 2-sided [-4.51 to 2.21] — Difference is calculated as BIIB033 100 mg/kg - placebo

5. Secondary Outcome: Change in SD-OCT Average RGCL/IPL at Week 24: Per-protocol Population
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 36 | 33
µm | -10.17 (1.29) | -11.93 (1.35)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; Test type: Superiority or Other; p = 0.3505, ANCOVA; Difference = -1.76, 95% CI 2-sided [-5.50 to 1.98]

6. Secondary Outcome: Change in Low-contrast Letter Acuity (LCLA) at Week 24: ITT Population
Description: Adjusted mean change in LCLA at Week 24 from baseline as determined by 1.25% and 2.5% low contrast Sloan letter charts, adjusted for the baseline LCLA value. The fellow eye is the reference eye for the inter-eye asymmetry. The range for LCLA assessment is 0-60.
Time Frame: Baseline, Week 24
Population: ITT population: all randomized subjects who received at least 1 dose of study treatment (BIIB033 or placebo) with an LCLA assessment at Baseline. LOCF imputation was used if Week 24 data were missing.
Measure: Mean (Standard Deviation); unit: letters on a chart
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 41 | 39
letters on a chart
  LCLA 1.25% chart | 8.1 (1.8) | 6.5 (1.9)
  LCLA 2.5% chart | 11.9 (2.0) | 11.0 (2.0)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; LCLA 1.25% chart; Test type: Superiority or Other; p = 0.5371, ANCOVA; Difference = -1.6, 95% CI 2-sided [-6.9 to 3.6] — Difference is calculated as BIIB033 100 mg/kg - placebo
Statistical Analysis 2: Comparison: Placebo vs BIIB033; LCLA 2.5% chart; Test type: Superiority or Other; p = 0.7741, ANCOVA; Difference = -0.8, 95% CI 2-sided [-6.5 to 4.9] — Difference is calculated as BIIB033 100 mg/kg - placebo

7. Secondary Outcome: Change in LCLA at Week 24: Per-protocol Population
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: letters on a chart
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 36 | 33
letters on a chart
  LCLA 1.25% chart | 7.2 (1.8) | 6.0 (2.0)
  LCLA 2.5% chart | 11.6 (2.0) | 10.8 (2.2)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; LCLA 1.25% chart; Test type: Superiority or Other; p = 0.6645, ANCOVA; Difference = -1.2, 95% CI 2-sided [-6.6 to 4.3]
Statistical Analysis 2: Comparison: Placebo vs BIIB033; LCLA 2.5%; Test type: Superiority or Other; p = 0.8015, ANCOVA; DIfference = -0.8, 95% CI 2-sided [-6.7 to 5.2]

8. Primary Outcome: Change in FF-VEP Latency at Week 24: Per-protocol Population
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Per-protocol Population: participants from the ITT population who completed the study, did not miss more than 1 dose of BIIB033 or placebo, and did not receive multiple sclerosis (MS)-modifying therapies during the study period, which were prohibited per protocol. LOCF imputation was used if Week 24 data were missing.
Measure: Mean (Standard Error); unit: msec
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 36 | 33
msec | 22.24 (2.61) | 14.69 (2.72)
Statistical Analysis 1: Comparison: Placebo vs BIIB033; Test type: Superiority or Other; p = 0.0504, ANCOVA; Difference = -7.55, 95% CI 2-sided [-15.12 to 0.01]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. An SAE was any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigators, placed the subject at immediate risk of death (a life-threatening event); however, this did not include an event that, had it occurred in a more severe form, might have caused death; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigators, could have jeopardized the subject or may have required intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: 32 weeks
Population: Safety population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | BIIB033
Number analyzed (Participants) | 41 | 41
participants
  Participants with an event | 34 | 34
  Participants with a moderate or severe event | 22 | 21
  Participants with a severe event | 2 | 3
  Participants with a related event | 8 | 14
  Participants with a serious event | 2 | 5
  Participants with a related serious event | 0 | 3
  Participants discontinuing treatment due to event | 1 | 3
  Participants withdrawing from study due to event | 2 | 3

10. Secondary Outcome: Summary of BIIB033 Concentration
Description: One pre-dose pharmacokinetic (PK) sample and 1 post-dose PK sample (approximately between 1 and 3 hours after the end of IV infusion) were collected for all participants on Day 1 and at Weeks 4 through 20 (every 4 weeks). Additionally, only 1 PK sample was collected at Week 24 and Week 32. (There was no dosing on Week 24 and Week 32, so only one blood sample for BIIB033 concentration was taken.) Samples collected at early termination visits were treated as predose samples for the next scheduled visit.
Time Frame: Up to 32 weeks
Population: PK analysis population: all participants who received at least 1 dose of BIIB033 and had at least 1 serum concentration data on record. n=number of participants with a sample at given timepoint.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | BIIB033
Number analyzed (Participants) | 41
µg/mL
  Baseline predose; n=41 | 0.00 [0.00 to 3.22]
  Baseline postdose; n=40 | 2030.00 [1370.00 to 3200.00]
  Week 4 predose; n=41 | 375.00 [14.60 to 2960.00]
  Week 4 postdose; n=37 | 2350.00 [368.00 to 3590.00]
  Week 8 predose; n=38 | 537.00 [32.70 to 1130.00]
  Week 8 postdose; n=36 | 2585.00 [550.00 to 4220.00]
  Week 12 predose; n=36 | 622.00 [39.90 to 3230.00]
  Week 12 postdose; n=34 | 2695.00 [542.00 to 4240.00]
  Week 16 predose; n=35 | 593.00 [173.00 to 1320.00]
  Week 16 postdose; n=34 | 2500.00 [1560.00 to 4590.00]
  Week 20 predose; n=37 | 673.00 [107.00 to 4760.00]
  Week 20 postdose; n=35 | 2530.00 [366.00 to 3990.00]
  Week 24; n=37 | 624.00 [4.30 to 1060.00]
  Week 32; n=33 | 82.70 [2.56 to 339.00]

ADVERSE EVENTS:
Time Frame: AEs were monitored from administration of first dose of study treatment through to Week 32 visit. SAEs were monitored from signing of the Informed Consent Form (ICF) through to Week 32 visit.
Groups:
- BIIB033 100 mg/kg: BIIB033 100 mg/kg via IV infusion once every 4 weeks for 20 weeks (a total of 6 doses)
Arm/Group | Placebo | BIIB033 100 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/41 | 5/41
Other Adverse Events (participants affected / at risk) | 25/41 | 27/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | BIIB033 100 mg/kg (N=41)
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Viral pericarditis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | BIIB033 100 mg/kg (N=41)
Colour blindness acquired (Eye disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 5 | 6
Influenza (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 13 | 12
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Dysaesthesia (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 11 | 11
Multiple sclerosis (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 4
Uhthoff's phenomenon (Nervous system disorders) | 6 | 3
Visual field defect (Nervous system disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.